CLINICAL TRIAL: NCT04998240
Title: A Phase 2, Observer-blind, Randomized Study to Assess the Safety and Immunogenicity of Heterologous Prime-boost COVID-19 Vaccines Regimens in Individuals Aged 18 to 65 Years in Mozambique and Madagascar.
Brief Title: Mix and Match Heterologous Prime-Boost Study Using Approved COVID-19 Vaccines
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Vaccine Institute (Other)
Collaborators: The Coalition for Epidemic Preparedness Innovations (CEPI) (Unknown); Instituto Nacional de Saúde, Mozambique (Other Government); University of Antananarivo (Unknown); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Harvard University (Other); Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IVI-ECOVA-02
Record Dates: First submitted 2021-07-29; First posted 2021-08-10 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Covid19
Keywords: SARS-CoV-2, Vaccines, Mix and Match Trial
MeSH Terms: conditions — COVID-19 | interventions — Ad26COVS1; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The primary analysis of this study will be a non-inferiority comparison between heterologous versus homologous boost arms 4 weeks after second vaccination within each group of the studied COVID-19 vaccines, i.e., the A1 arm (BBIBP-CorV, Ad26.COV2.S) will be compared with the A2 arm (BBIBP-CorV, BBIBP-CorV), and the B1 arm (Ad26.COV2.S, BBIBP-CorV) will be compared with the B2 arm (Placebo, Ad26.COV2.S). All 360 participants will be used for the primary analysis and the secondary analysis.
Who Masked: Outcomes Assessor
Masking Description: This is an observer-blind study. So in this study only the outcome assessors should be blinded namely the clinical staff in charge of the clinical outcomes assessment and the laboratory analysts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prime BBIBP-CorV, Boost Ad26.COV2.S (A1) (Experimental): The randomized study participants will receive Prime BBIBP-CorV vaccine followed by Booster dose of Ad26.COV2.S vaccine (A1).
  Interventions: Biological: BBIBP-CorV - Inactivated SARS-CoV-2 vaccine (Vero cell); Biological: Ad26.COV2.S (Recombinant, replication-incompetent adenovirus serotype 26 (Ad26) vector encoding a full-length and stabilized SARS-CoV-2 spike protein),
- Prime BBIBP-CorV, Boost BBIBP-CorV (A2) (Experimental): The randomized study participants will receive Prime BBIBP-CorV vaccine followed by Booster dose of BBIBP-CorV vaccine (A2).
  Interventions: Biological: BBIBP-CorV - Inactivated SARS-CoV-2 vaccine (Vero cell)
- Prime Ad26.COV2.S, Boost BBIBP-CorV (B1) (Experimental): The randomized study participants will receive Prime Ad26.COV2.S vaccine followed by Booster dose of BBIBP-CorV vaccine (B1).
  Interventions: Biological: BBIBP-CorV - Inactivated SARS-CoV-2 vaccine (Vero cell); Biological: Ad26.COV2.S (Recombinant, replication-incompetent adenovirus serotype 26 (Ad26) vector encoding a full-length and stabilized SARS-CoV-2 spike protein),
- Prime Placebo, Boost Ad26.COV2.S (B2) (Experimental): The randomized study participants will receive Prime Placebo vaccine followed by Booster dose of Ad26.COV2.S (B2).
  Interventions: Biological: Ad26.COV2.S (Recombinant, replication-incompetent adenovirus serotype 26 (Ad26) vector encoding a full-length and stabilized SARS-CoV-2 spike protein),; Biological: Placebo - Normal saline (0.9% sodium chloride solution)

INTERVENTIONS:
Biological: BBIBP-CorV - Inactivated SARS-CoV-2 vaccine (Vero cell) — The Inactivated SARS-CoV-2 vaccine (Vero cell)- BBIBP-CorV manufactured by Beijing Institute of Biological Products (BIBP), China National Biotec Group (CNBG), Sinopharm, Beijing, People's Republic of China
  Dose formulation: A liquid formulation containing 4μg total protein with aluminum hydroxide adjuvant (0·45 mg/mL) per 0·5 mL (2-dose schedule followed by a booster dose).
  Mode of Administration:
  Intramuscular
  Storage Conditions: 2°C to 8°C
  Arms: Prime Ad26.COV2.S, Boost BBIBP-CorV (B1); Prime BBIBP-CorV, Boost Ad26.COV2.S (A1); Prime BBIBP-CorV, Boost BBIBP-CorV (A2)
Biological: Ad26.COV2.S (Recombinant, replication-incompetent adenovirus serotype 26 (Ad26) vector encoding a full-length and stabilized SARS-CoV-2 spike protein), — Ad26.COV2.S (Recombinant, replication-incompetent adenovirus serotype 26 (Ad26) vector encoding a full-length and stabilized SARS-CoV-2 spike protein), manufactured by Johnson and Johnson in the United States of America.
  Dose formulation: One dose (0.5 ml) contains contains 5 x 10 10 virus particles
  Mode of administration: Intramuscular
  Storage Conditions: 2°C to 8°C
  Arms: Prime Ad26.COV2.S, Boost BBIBP-CorV (B1); Prime BBIBP-CorV, Boost Ad26.COV2.S (A1); Prime Placebo, Boost Ad26.COV2.S (B2)
Biological: Placebo - Normal saline (0.9% sodium chloride solution) — Placebo - Normal saline (0.9% sodium chloride solution)
  Dose formulation: Not Applicable
  Mode of administration: Intramuscular
  Storage conditions: 15°C to 30°C
  Arms: Prime Placebo, Boost Ad26.COV2.S (B2)

SUMMARY:
This is an observer-blind, randomized study which aims to assess the immune response and the safety of two different approved vaccines for first and second dose in healthy adults.

DETAILED DESCRIPTION:
This is a phase 2, observer-blind, randomized study to assess the safety and the immunogenicity of heterologous prime-boost COVID-19 vaccines regimens in healthy adults aged 18 to 65 years using two approved vaccines (Sinopharm / CNBG Vaccine (BBIBP-CorV) and Johnson & Johnson Vaccine (Ad26.COV2.S)).

The study will consist of 2 cohorts, one for main immunology endpoints (N=260, 65 per study arm) and one for more detailed immunological assessment (N=100, 25 per study arm). Two doses of vaccine will be administered intramuscularly 4 week apart. All the study participants will be follow-up for 12 months from the administration of first vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 65 years old at the time of consent.
* Residing within the area of the study and planning to stay for the study duration.
* HIV negative test result on the day of screening (for those who do not have a documented HIV test results in the last three months of screening).
* Female volunteers of childbearing potential with a negative pregnancy test on the day(s) of screening and vaccination, practicing/willing to practice continuous effective contraception* recommended by the National Health System up to 12 weeks after the booster vaccination..
* Agreement to refrain from blood donation during the course of the study.
* Able and willing to comply with all study requirements, based on the assessment of the investigator.
* Willingness to provide written informed consent before any trial procedure * Effective contraception is defined as follows: contraceptive medications delivered orally, intramuscularly, vaginally, or implanted underneath the skin, surgical methods (hysterectomy or bilateral tubal ligation), condoms, diaphragms, intrauterine device (IUD), and abstinence.

Exclusion Criteria:

* Pregnancy, lactation, or intention to become pregnant during the vaccination phase through three months after the booster dose.
* Prior receipt/ planned receipt of any vaccine other than the study intervention within 28 days before and after each study vaccination.
* Previous participation in any COVID-19 vaccination trial or vaccination campaign.
* Administration of immunoglobulins and/ or any blood products within the three months preceding the administration of the study vaccine.
* Known infection with hepatitis B, C virus.
* Known history of allergy or anaphylaxis to study vaccine components and/or excipients or other medications, or any other allergies deemed by the investigator to increase the risk of an adverse reaction.
* History of bleeding disorder (e.g., factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
* Continuous use of the anticoagulants, such as coumarins and related anticoagulants.
* Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, renal disease, liver disease, endocrine disorders, and neurological illness (mild/moderate well controlled comorbidities are allowed).
* Any clinically significant abnormal finding on screening as judged by the investigator.
* Confirmed SARS-CoV-2 infection at enrollment.
* Any confirmed or suspected immunosuppressive or immunodeficient state, asplenia, recurrent severe infections and chronic use (more than 14 days) immunosuppressant medication within 3 months prior to recruitment (topical steroids are allowed).
* Any other finding which in the opinion of the investigators would increase the risk of an adverse outcome from participation in the trial or result in incomplete or poor-quality data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titers (GMTs) of anti-SARS-CoV-2 neutralizing antibodies | Four Weeks after second dose
  Geometric Mean Titers (GMTs) of anti-SARS-CoV-2 neutralizing antibodies using a neutralization assay four weeks after the second dose, in COVID-19 seronegative participants following immunization with heterologous and homologous prime-boost COVID-19 vaccines regimens.
Incidence of SAEs and AESI observed at any time point during the entire study period | Till 12 months follow-up visit
  Incidence of SAEs and AESI observed at any time point during the entire study period, among all study participants of heterologous and homologous prime-boost COVID-19 vaccines regimens
Incidence of solicited reactions within 7 days (local reactions) and 14 days (systemic reactions) | Within 7 days (local reactions) and 14 days (systemic reactions) following each vaccination
  Incidence of solicited reactions within 7 days (local reactions) and 14 days (systemic reactions) following each vaccination in all study participants of heterologous and homologous prime-boost COVID-19 vaccines regimens.
Incidence of unsolicited adverse events that are within 28 days after each vaccination | Within 28 days after each vaccination
  Incidence of unsolicited adverse events that are within 28 days after each vaccination in all study participants of heterologous and homologous prime-boost COVID-19 vaccines regimens.
Incidence of changes in laboratory safety measures from baseline to day 28 after each vaccination | Within 28 days after each vaccination
  Incidence of changes in laboratory safety measures from baseline to day 28 after each vaccination, in all study participants of heterologous and homologous prime-boost COVID-19 vaccines regimens

SECONDARY OUTCOMES:
Geometric Mean Titers (GMTs) and Geometric Mean Fold Rise (GMFR) | Till 12 months follow-up visit
  * GMTs of anti-SARS-CoV-2 neutralizing antibodies as measured by neutralization assay at Day 0, Day 28, Day 196, Day 364
  * GMFR from baseline of anti-SARS-CoV-2 neutralizing antibodies as measured by neutralization assay at Day 0, Day 28, Day 196, Day 364
  * Percentage of participants achieving 4-fold or more rise from baseline of anti-SARS-CoV-2 neutralizing antibodies as measured by neutralization assay at Day 0, Day 28, Day 196, Day 364
Geometric Mean Titers (GMTs) and Geometric Mean Fold Rise (GMFR) | Till 12 months follow-up visit
  * GMTs of anti-SARS-CoV-2 anti-spike IgG as measured by immunoassay, anti-SARS-CoV-2 pseudoneutralizing antibodies as measured by pseudo-neutralization assay, and anti-SARS-CoV-2 anti-nucleocapsid IgG at Day 0, Day 28, Day 56, Day 196, Day 364
  * GMFR from baseline of anti-SARS-CoV-2 anti-spike IgG as measured by immunoassay, anti-SARS-CoV-2 pseudo-neutralizing antibodies as measured by pseudo-neutralization assay, and anti-SARS-CoV-2 anti-nucleocapsid IgG at Day 0, Day 28, Day 56, Day 196, Day 364
  * Percentage of participants achieving 4-fold or more rise from baseline for anti-SARS-CoV-2 anti-spike IgG as measured by immunoassay, anti-SARS-CoV-2 pseudoneutralizing antibodies as measured by pseudo-neutralization assay, and anti-SARS-CoV-2 anti-nucleocapsid IgG at Day 0, Day 28, Day 56, Day 196, Day 364

OTHER OUTCOMES:
Cellular immune responses against SARS-CoV-2 | Till 12 months follow-up visit
  Cellular immune responses against SARS-CoV-2 by ELISpot and by Intracellular Cytokine Staining (ICS) (Th1/Th2) at days 0, 14, 28, 42, 56, 196, 364, following immunization with heterologous and homologous prime-boost COVID-19 vaccines regimens, in the participants of immunology cohort.
GMTs, GMFR from baseline | Till 12 months follow-up visit
  * GMTs of anti-SARS-CoV-2 anti-spike IgG, anti-nucleocapsid IgG against SARS-CoV-2, nAbs and pnAbs against SARS-CoV-2, cellular immune response against SARS-CoV-2, post prime or boost dose, and within one week in all participants being found to be SARS-CoV-2 positive by testing.
  * GMFR from baseline of anti-SARS-CoV-2 anti-spike IgG, anti-nucleocapsid IgG against SARS-CoV-2, nAbs and pnAbs against SARS-CoV-2, cellular immune response against SARS-CoV-2, post prime or boost dose, and within one week in all participants being found to be SARS-CoV-2 positive by testing.
  * Percentage of participants achieving 4-fold or more rise from baseline for anti-SARS-CoV-2 anti-spike IgG, anti-nucleocapsid IgG against SARS-CoV-2, nAbs and pnAbs against SARS-CoV-2, cellular immune response against SARS-CoV-2, post prime or boost dose, and within one week in all participants being found to be SARS-CoV-2 positive by testing.
Genome sequencing of SARS-CoV-2 viruses isolated post prime or booster dose | After diagnosis of SARS-CoV-2 infection
  Genome sequencing of SARS-CoV-2 viruses isolated post prime or boost, after diagnosis of SARS-CoV-2 infection, in all study participants of heterologous and homologous prime-boost COVID-19 vaccines regimens
Profile of vaccine-induced humoral response against SARS-CoV-2 | Till 12 months follow-up visit
  Profile of vaccine-induced humoral response against SARS-CoV-2 using systems serology at days 0, 14, 28, 42, 56, 196, 364, in study participants of immunology subset cohort, following immunization with heterologous and homologous prime-boost COVID-19 vaccines regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Marks, PhD, Principal Investigator — International Vaccine Institute; Ilesh Jani, PhD, Principal Investigator — Instituto Nacional de Saúde, Mozambique; Raphael Rakotozandrindrainy, MD, Principal Investigator — Madagascar Institute for Vaccine Research (MIVR), University of Antananarivo
Locations (2):
- Madagascar Institute for Vaccine Research (MIVR), University of Antananarivo, Antananarivo, Madagascar
- Centro de Investigação e Treino em Saúde da Polana Caniço - Instituto Nacional de Saúde, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ramgi P, Siribie M, Rakotozandrindrainy N, Bule O, Shrivastava H, Chambule L, Park EL, Fernando C, Boque J, Macuiana R, Razafimanantsoa R, Rakotozandrindrainy N, Razafindrabe TJL, Rakotoarisoa AN, Raminosoa TM, Derandrainy HL, Rakotoson MM, de Silva CSS, Mutombene M, Massinga C, Langa JP, Guarnacci T, Kang SSY, Jo SK, Jeon HJ, Excler JL, Yang Y, Wang S, Sugimoto JD, Yang JS, Shim BS, Binger T, Capitine IU, Aziz AB, Park JY, Kim DR, Rakotozandrindrainy R, Jani IV, Tadesse BT, Marks F. Immunogenicity and Safety of Heterologous Versus Homologous Prime-Boost Regimens With BBIBP-CorV and Ad26.COV2.S COVID-19 Vaccines: A Multicentric, Randomized, Observer-Blinded Non-inferiority Trial in Madagascar and Mozambique. Clin Infect Dis. 2025 Jul 22;80(Supplement_1):S37-S46. doi: 10.1093/cid/ciaf130. PMID 40694514
- See also: Description Mozambique COVID-19 Situation — https://covid19.who.int/region/afro/country/mz